CLINICAL TRIAL: NCT05258942
Title: MyLeukoMAP™ Genomic Survival Prediction Assay for Heart Failure Pivotal Clinical Study
Brief Title: MyLeukoMAP™ Genomic Survival Prediction Assay Pivotal Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LeukoLifeDx Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: LLDx1012021
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Heart Failure Patients Scheduled for Coronary Artery Bypass Graft (CABG) Surgery: Heart Failure Patients Scheduled for Coronary Artery Bypass Graft (CABG) Surgery
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Percutaneous Coronary Interventions (PCI): Heart Failure Patients Scheduled for Percutaneous Coronary Interventions (PCI)
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Aortic Valve Replacement (AVR) Surgery: Heart Failure Patients Scheduled for Aortic Valve Replacement (AVR) Surgery
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Mitral Valve Replacement (MVR) Surgery: Heart Failure Patients Scheduled for Mitral Valve Replacement (MVR) Surgery
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Transcatheter Aortic Valve Replacement (TAVR): Heart Failure Patients Scheduled for Transcatheter Aortic Valve Replacement (TAVR)
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Transcatheter Mitra Clip: Heart Failure Patients Scheduled for Transcatheter Mitra Clip
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Ventricular Tachycardia Ablation: Heart Failure Patients Scheduled for Ventricular Tachycardia Ablation
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Stellate Gangliectomy: Heart Failure Patients Scheduled for Stellate Gangliectomy
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Mechanical Circulatory Support (MCS) Surgery: Heart Failure Patients Scheduled for Mechanical Circulatory Support (MCS) Surgery
  Interventions: Other: Observational
- Heart Failure Patients Scheduled for Heart Transplantation (HTx) Surgery: Heart Failure Patients Scheduled for Heart Transplantation (HTx) Surgery
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Blood samples will be collected within 30 days before scheduled surgical / interventional therapy for Heart Failure. The study will not impact patient treatment in any way.

SUMMARY:
The MyLeukoMAP™ Pivotal Clinical Study will assess the accuracy of MyLeukoMAP™, a new molecular blood test, performed within 30 days before scheduled surgical / interventional therapies for Heart Failure, to determine its effectiveness in improving clinical decision support by providing a quantitative prediction of low, indeterminate, or high risk of death one year after surgical / interventional therapies that is not identified by current diagnostic tools.

DETAILED DESCRIPTION:
The MyLeukoMAP™ Pivotal Clinical Study will assess the accuracy of MyLeukoMAP™, a new molecular blood test, performed within 30 days before scheduled surgical / interventional therapies for Heart Failure, to determine its effectiveness in improving clinical decision support by providing a quantitative prediction of low, indeterminate, or high risk of death one year after surgical / interventional therapies that is not identified by current diagnostic tools.

Patients scheduled for one of 10 different Heart Failure surgical / interventional therapies will be identified and consented. Four clinical parameters will be collected for each patient: age, white blood cell count, blood pressure, and respiratory rate. Blood samples will be collected concurrent with a routine preoperative blood draw, and peripheral blood mononuclear cells (PBMC's) will be isolated. The PBMC samples will be shipped to ResearchDx, Irvine, CA, for testing using the MyLeukoMAP™ genomic survival prediction assay. Patient 1-year postoperative survival/non-survival data will be reported for each patient.

The samples will be tested 1-year after the intervention of the last enrolled patient, and the data will be compared to actual patient 1-year survival to determine the survival prediction accuracy of the assay. The investigators anticipate that the assay will better identify those 20% of patients who currently do not achieve 1-year postoperative survival, and who would have better odds of survival by remaining on medical therapy, but who cannot be identified with current tools.

ELIGIBILITY:
Inclusion Criteria:

Criteria #1: AdHF with NYHA III/IV

Criteria #2: Left Ventricular Ejection Fraction (LVEF) <35% or >2+valvular disease severity & >low risk Society of Thoracic Surgeons (STS)-score

Criteria #3: Evaluation for interventions including CABG/PCI (Stratum #1, Ischemia), Surgical Valve Replacement/TAVR/Mitra-Clip (Stratum #2, Overload), VT-Ablation/Stellate Gangliectomy (Stratum #3, Arrhythmia), or MCS/HTx (Stratum #4, Contractility)

-

Exclusion Criteria:

Criteria #1: No informed consent Criteria #2: <18 years old

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study Participants: All study participants will be referred to the AdHF Program at one of the study investigational sites, evaluated for the various therapeutic options outlined below, and scheduled for HF-surgical / interventional therapy. All patients will be optimized regarding HF therapy, consented, and prescribed one of 10 HF procedures according to established guidelines, based on the recommendations of the AdHF team of the participating study centers.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Survival / Non-Survival | 1-year (365-455 Days) Post Intervention
  Patient Survival Status

CONTACTS AND LOCATIONS:
Overall Officials: Megan Kamath, MD, Principal Investigator — University California Los Angeles
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - AdventHealth Orlando, Orlando, Florida
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bondar G, Togashi R, Cadeiras M, Schaenman J, Cheng RK, Masukawa L, Hai J, Bao TM, Chu D, Chang E, Bakir M, Kupiec-Weglinski S, Groysberg V, Grogan T, Meltzer J, Kwon M, Rossetti M, Elashoff D, Reed E, Ping PP, Deng MC. Association between preoperative peripheral blood mononuclear cell gene expression profiles, early postoperative organ function recovery potential and long-term survival in advanced heart failure patients undergoing mechanical circulatory support. PLoS One. 2017 Dec 13;12(12):e0189420. doi: 10.1371/journal.pone.0189420. eCollection 2017. PMID 29236770
- [Result] Deng MC. A peripheral blood transcriptome biomarker test to diagnose functional recovery potential in advanced heart failure. Biomark Med. 2018 Jun;12(6):619-635. doi: 10.2217/bmm-2018-0097. Epub 2018 May 8. PMID 29737882
- [Result] Bondar G, Cadeiras M, Wisniewski N, Maque J, Chittoor J, Chang E, Bakir M, Starling C, Shahzad K, Ping P, Reed E, Deng M. Comparison of whole blood and peripheral blood mononuclear cell gene expression for evaluation of the perioperative inflammatory response in patients with advanced heart failure. PLoS One. 2014 Dec 17;9(12):e115097. doi: 10.1371/journal.pone.0115097. eCollection 2014. PMID 25517110